CLINICAL TRIAL: NCT04539509
Title: The Effects of Early Prescribed Aerobic Exercise on Recovery and Post-concussive Symptoms in Adults
Brief Title: Post-Concussion Aerobic Exercise
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Revising study protocol.
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-5899; 15-9214 (Other: University Health Network REB - Legacy ID)
Record Dates: First submitted 2020-08-19; First posted 2020-09-07 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2022-11

CONDITIONS: Concussion, Mild; Mild Traumatic Brain Injury
Keywords: Concussion; Mild traumatic brain injury; Aerobic exercise
MeSH Terms: conditions — Brain Concussion | interventions — Exercise Test

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The primary outcome (recovery) is determined using a 3 step approach. Each assessor responsible for one of the three steps, will be blind to at least ONE other recovery determinant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Monitoring (Active Comparator): Participants will be given a heart rate monitor to wear on their wrist for the duration of the study (i.e. until recovered, or 8 weeks post-injury, whatever comes first).
  Interventions: Device: Monitoring
- Monitoring + Treadmill Test (Placebo Comparator): In addition to wearing the heart rate monitor, participants will undergo a treadmill test at each appointment.
  Interventions: Behavioral: Treadmill Test; Device: Monitoring
- Monitoring + Treadmill Test + Specific Exercise Prescription (Experimental): In addition to wearing the heart rate monitor, and completing a treadmill test at each appointment, participants will receive an exercise prescription based on the results of the treadmill test. They will be prescribed 30 minutes of structured aerobic exercise, 5 times per week, at a heart rate determined by their treadmill test.
  Interventions: Behavioral: Exercise Prescription; Behavioral: Treadmill Test; Device: Monitoring

INTERVENTIONS:
Behavioral: Exercise Prescription — A specific exercise prescription, based on the results of a treadmill test.
  Arms: Monitoring + Treadmill Test + Specific Exercise Prescription
Behavioral: Treadmill Test — A symptom-limited treadmill test, using the Buffalo Concussion Treadmill Test (BCTT) protocol.
  Arms: Monitoring + Treadmill Test; Monitoring + Treadmill Test + Specific Exercise Prescription
Device: Monitoring — Activity monitoring using a Fitbit.

SUMMARY:
This study is looking at the specific role of an exercise prescription on recovery from concussion symptoms in the general population.

DETAILED DESCRIPTION:
435 people will participate in this study.

A physician will review a participant's medical history to determine if physical activity is appropriate for them. They will then be randomly assigned to 1 of 3 study groups:

1. Monitoring- participants will be given a heart rate monitor to wear on their wrist for the duration of the study (until "recovered", or until 8 weeks post-concussion, whatever comes first).
2. Monitoring + Treadmill Testing- in addition to wearing the heart rate monitor, they will undergo a treadmill test at each appointment.
3. Monitoring + Treadmill Testing + Specific Exercise Prescription- in addition to wearing the heart rate monitor, and treadmill test, they will receive an exercise prescription based on the results of the treadmill test.

The randomization is by chance. Participants have a 40/20/40% respective chance of being assigned to the study groups above. This means that out of every 5 people: 2 people will be assigned to the group 1, 1 will be assigned to the group 2, and 2 will be assigned to the group 3. Both participants and the study doctor will be aware which group participants are in.

Regardless of the group assigned, participants will receive an exercise prescription form at each appointment, as per usual care. The prescription will be based on the physician's judgement. If a participant is in group 3, their prescription will also take into account the results of the treadmill test.

Recovery will be determined using a 3-step approach:

1. Self-reported symptoms,
2. Clinic physician's opinion,
3. Treadmill test results (if applicable).

ELIGIBILITY:
Inclusion Criteria:

* Patients that provide written informed consent prior to entry into the study
* Patients referred from the emergency department (ED) with recent (<1 week) diagnosis of concussion by ED physician
* GCS score of 13-15 on presentation to the ED
* SCAT score > 9 at week 1
* Physician cleared for exercise; low risk for cardiac disease (defined as no cardiopulmonary symptoms and meet no more than one risk factor for heart disease)
* Willing to exercise

Exclusion Criteria:

* Evidence of intracranial hemorrhage, contusion or injury on brain imaging (CT Scan)
* Beta-blocker medication
* High dose (>50mg/day) tricyclic antidepressant medication
* Pre-existing or current orthopedic injuries preventing exercise
* Pre-existing vestibular disease preventing exercise
* Heartrate increase <30 bpm from rest on treadmill test
* Deemed asymptomatic from concussion by clinic physician
* Unable/unwilling to follow commands

Ages: 17 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Recovered | Assessed at week 8 post-concussion.
  "Recovery" (yes/no) will be determined using a 3-step approach:
  1. Self-reported symptoms (using the Sport Concussion Assessment Tool [SCAT], Symptom Inventory),
  2. Clinic physician's opinion,
  3. Treadmill test results (if applicable).

SECONDARY OUTCOMES:
Percentage of Participants Recovered | Assessed at week 2 post-concussion.
Percentage of Participants Recovered | Assessed at week 4 post-concussion.
Percentage of Participants who have Returned to Work/School | Assessed at week 2 post-concussion.
  Time at which participants return to part-time and/or full-time work or school activities.
Percentage of Participants who have Returned to Work/School | Assessed at week 4 post-concussion.
Percentage of Participants who have Returned to Work/School | Assessed at week 8 post-concussion.
Brief Symptom Inventory-18 (BSI-18) Global Severity Index Score | Assessed at week 2 post-concussion.
  Measured using the Brief Symptom Inventory (BSI)-18. Global scores, as well as somatization, depression, and anxiety sub-scales will be included.
  Global scores are calculated by adding up participants self-reported score (0-72), with high scores indicating more psychological distress. These scores are then compared to gender-stratified norms. Sub-scales are scored on a 0-24 scale, again higher scores indicating more psychological distress (sub-scales also compared to gender-stratified norms).
Brief Symptom Inventory-18 (BSI-18) Global Severity Index Score | Assessed at week 4 post-concussion.
Brief Symptom Inventory-18 (BSI-18) Global Severity Index Score | Assessed at week 8 post-concussion.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bayley, MD, Principal Investigator — University Health Network, Toronto Rehabilitation Institute
Locations (1):
- Toronto Rehabilitation Institute - University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No IDP sharing plan.

REFERENCES:
- [Background] Haider MN, Leddy JJ, Wilber CG, Viera KB, Bezherano I, Wilkins KJ, Miecznikowski JC, Willer BS. The Predictive Capacity of the Buffalo Concussion Treadmill Test After Sport-Related Concussion in Adolescents. Front Neurol. 2019 Apr 24;10:395. doi: 10.3389/fneur.2019.00395. eCollection 2019. PMID 31105634
- [Background] Lawrence DW, Richards D, Comper P, Hutchison MG. Earlier time to aerobic exercise is associated with faster recovery following acute sport concussion. PLoS One. 2018 Apr 18;13(4):e0196062. doi: 10.1371/journal.pone.0196062. eCollection 2018. PMID 29668716
- [Background] Leddy JJ, Willer B. Use of graded exercise testing in concussion and return-to-activity management. Curr Sports Med Rep. 2013 Nov-Dec;12(6):370-6. doi: 10.1249/JSR.0000000000000008. PMID 24225521